CLINICAL TRIAL: NCT04614740
Title: Single-arm, Open, Multi-center Phase I/Phase II Clinical Study to Assess the Safety, Tolerability, Pharmacokinetic and Effectiveness of VC004
Brief Title: The Phase I/Phase II Clinical Study of VC004 in Patients With Localized Advanced/Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VC004-101
Record Dates: First submitted 2020-10-12; First posted 2020-11-04 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-10

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: Safety, Tolerability, Pharmacokinetic, Effectiveness
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Single arm clinical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VC004 (Experimental): 1. Dose escalation stage: subjects in the 50 mg, 100 mg, 200 mg, and 300 mg dose groups took a single oral dose on the first day; starting from the fourth day, each group of subjects took the corresponding dose twice a day. 2. Dose expansion stage: subjects in the 100mg and 200mg dose groups took the corresponding dose twice a day on an empty stomach; 3. Phase II clinical trial stage: oral administration twice a day before meals, and the dosage is to be determined.
  Interventions: Drug: VC004

INTERVENTIONS:
Drug: VC004 — 25 mg capsules,50 mg capsules,100 mg capsules.

SUMMARY:
Dose-escalation study will be conducted in patients with locally advanced/metastatic solid tumors who have failed standard treatment, or cannot tolerate standard treatment, or have no recommended standard treatment, or do not apply standard treatment, to evaluate the safety, PK, tolerability and effectiveness of VC004. According to the efficacy, safety and PK of dose-escalation study , the investigator and the sponsor jointly determine the dose for dose extension, and evaluate the anti-tumor effect of VC004 on NTRK fusion-positive subjects, and provide more information for RP2D.

According to the tolerability and pharmacokinetic results of dose-escalation study , an appropriate dose or MTD will be selected, namely RP2D, to further assess anti-tumor efficacy and safety in patients with NTRK fusion-positive locally advanced/metastatic solid tumors . ORR will be chosen as the main efficacy indicator to evaluate the anti-tumor efficacy and safety of VC004 .

ELIGIBILITY:
Inclusion Criteria:

* All subjects or legal representatives are willing and able to sign ICF approved by the ethics committee before starting any screening procedures；
* Male or female, age ≥18 years old
* Patients with locally advanced or metastatic solid tumors diagnosed by histology or cytology, or currently have no standard treatment, have failed the standard treatment, or are intolerant to the standard treatment or are not suitable for the standard treatment at this stage。 The first part of the dose escalation stage: locally advanced or metastatic solid tumors, including but not limited to salivary gland cancer, thyroid cancer, soft tissue sarcoma, liposarcoma, etc.
* Subject's baseline lesion requirements: According to the definition of RECIST v1.1 or RANO, the subject must have at least one measurable lesion (applicable to NTRK fusion-positive locally advanced or metastatic solid tumors)。
* Subjects with primary central nervous system (CNS) tumors must meet the following criteria (only the first part of the dose expansion phase and the second part are applicable)

  * According to the guidelines or CNS tumor type, have received treatment including radiotherapy and/or chemotherapy, and the interval between radiotherapy and the first treatment with study drug is at least 12 weeks.
  * According to the definition of RANO, there is at least one measurable lesion in magnetic resonance imaging (MRI), which can be visualized on ≥2 axial films with a thickness of 5 mm, and the longitudinal diameters perpendicular to each other are> 10 mm.
  * The imaging examination was performed within 28 days before enrollment. If you receive glucocorticoid treatment, a stable dose of glucocorticoid is required at least 5 days before imaging evaluation.
* The Eastern Cooperative Oncology Group (ECOG) score is ≤2 points (0-1 points are required for the dose-escalation stage)
* The estimated survival time is ≥12 weeks.
* The subject must have appropriate organ and hematological functions (have not received blood transfusion, EPO, G-CSF or other medical supportive treatment within 14 days before the administration of the study drug)。
* Premenopausal women who are likely to have children must have a pregnancy test within 7 days before starting treatment. The pregnancy test must be negative and must be non-lactating; Infertile women may not undergo pregnancy tests and contraception, but they must meet the following requirements: age 50 years or older, not using hormone therapy and menopause for at least 12 months, or have undergone sterilization. All enrolled patients (whether male or female) should take adequate contraceptive measures throughout the treatment period and 180 days after the end of treatment.

Exclusion Criteria:

* Patients have previously received any of the following treatments:

  * Patients have used any cytotoxic chemotherapeutic agents, targeted therapies, immunotherapies, or other anti-cancer drugs in the previous regimen within 4 weeks before the first administration ( e.g.Nitrosourea or mitomycin C for 6 weeks prior to first use of study drug, Oral fluorouracil and small-molecule targeted drugs are administered 2 weeks prior to the first use of the study drug or within 5 half-lives of the drug, whichever is longer.).
  * The time from receiving other experimental drugs or analogues to the first dose does not exceed the drug's 5 half-life or 14 days (whichever is longer).
  * Patients have used chinese herbal medicines and chinese herbal preparations with antitumor as an indication, chinese herbal medicines and chinese herbal preparations with tumor adjuvant therapeutic effect within 14 days before the first administration.
* Patients have undergone major surgery within 4 weeks prior to the first dose or are expected to undergo major surgery during the trial (excluding vascular access establishment procedures, biopsy procedures)
* Adverse reactions caused by previous treatment have not recovered to ≤1 grade (the dose-escalation stage does not include ≤2 grade hair loss, and the dose expansion stage and phase II clinical trials are comprehensively evaluated by the investigator).
* Primary central nervous system malignancy (only the first part of the dose escalation phase).
* Patients are known to have symptomatic or untreated brain metastases or other central nervous system metastases.CNS lesions that remain stable or show improvement after treatment with complete resection and/or radiation therapy are excluded, but require no glucocorticoids to control neurological symptoms within 14 days prior to entry into this study.
* There is any clinical basis suggesting a severe or uncontrolled systemic disease for which the investigator believes the patient is unsuitable for trial participation or which would affect the patient's compliance with the study protocol, such as stable or decompensated respiratory disease, cerebrovascular disease, liver disease, renal disease, uncontrolled diabetes, aortic dissection, aortic aneurysm, active bleeding-prone body, or those requiring systemic anti-infective therapy.
* Any clinically serious gastrointestinal abnormality that may affect the ingestion, transit, or absorption of study drugs.
* Patients have clinically significant cardiovascular diseases, including：

  * Left ventricular ejection fraction (LVEF) ≤ 50% by echocardiography during the screening period
  * Heart Failure, New York Heart Association (NYHA) grade III and above
  * Poorly controlled hypertension (BP ≥ 150/100 mmHg despite use of optimal therapy)
  * Past or current cardiomyopathy
  * Patients with atrial fibrillation and severe arrhythmia with ventricular rate> 100 bpm
  * Unstable ischemic heart disease (myocardial infarction (MI) within 6 months prior to starting study treatment, or angina that requires >1 nitrate per week to control symptoms)
* QTcF interval ≥450ms for males and ≥470ms for females (Fredericka formula: QTcF = QT/RR0.33)
* Patients had been treated with a strong CYP3A inhibitor or inducer within 7 days prior to the first administration of the study drug.
* Currently existing hepatitis B (hepatitis B surface antigen [HbsAg] positive or core antibody [HbcAb] positive and HBV DNA positive), hepatitis C (HCV anti-positive and HCV RNA positive), human immunodeficiency virus (HIV) infection and syphilis infection.
* Patients whom the investigators determine are not suitable for participation in the study for other reasons.
* Subjects are unwilling or unable to follow the protocol process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety&Tolerability | 4 years
  Adverse events (CTCAE5.0)and/or laboratory testsand/or electrocardiogramand/or echocardiogramand/or vital signsand/or physical examination
Phase II recommended dose(RP2D) | 1.5 years
  According to the tolerability and pharmacokinetic results of different dose groups completed during the dose escalation phase, an appropriate dose or MTD is selected as RP2D
Maximum tolerated dose(MTD)(If any) | 1.5 years
  If ≥2 cases of DLT are observed at a certain dose (up to 6 subjects), the dose will be considered an intolerable dose, and the previous dose group will be regarded as MTD
Objective response rate(ORR) | 4 years
  The proportion of subjects whose best overall response is CR or PR in the study assessed by IRC/investigator according to RECIST v1.1 or RANO

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0 min ，15 min，30 min，1 hour (h)，2 h，3 h，4 h，6 h，8 h，12 h，24 h，48 h
Peak time(Tmax) | 0 min ，15 min，30 min，1 hour (h)，2 h，3 h，4 h，6 h，8 h，12 h，24 h，48 h
half-time（t1/2） | 0 min ，15 min，30 min，1 hour (h)，2 h，3 h，4 h，6 h，8 h，12 h，24 h，48 h
Area Under the Curve From Time Zero to Last Quantifiable Concentration(AUC） | 0 min ，15 min，30 min，1 hour (h)，2 h，3 h，4 h，6 h，8 h，12 h，24 h，48 h
Apparent volume of distribution(Vz/F) | 0 min ，15 min，30 min，1 hour (h)，2 h，3 h，4 h，6 h，8 h，12 h，24 h，48 h
Duration of Remission (DOR) | 2.5 years
  Time from the first recording of remission (CR or PR) to the first recording of disease progression or death (whichever occurs first)
Progression-free survival (PFS) | 2.5 years
  The time from the subject receiving the first study treatment to the appearance of disease progression or death from any cause (whichever occurs first)
Overall survival (OS) | 2.5years
  The time from the date of first medication to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: yuankai shi, Principal Investigator — Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (21):
- China (21):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Hainan Cancer Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical Univercity Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Tianjin Cancer Hospital, Tianjin
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Hubei Cancer Hospital, Wuhan